CLINICAL TRIAL: NCT00061906
Title: Phase II Study Of Celecoxib In Metastatic Differentiated Thyroid Carcinoma
Brief Title: Celecoxib in Treating Patients With Progressive Metastatic Differentiated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Manisha Shah, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0239
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Head and Neck Cancer
Keywords: insular thyroid cancer; recurrent thyroid cancer; stage II follicular thyroid cancer; stage II papillary thyroid cancer; stage IV follicular thyroid cancer; stage IV papillary thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib — Treatment will be administered on an outpatient basis. Oral celecoxib will be given at the dose of 400 mg BID for total of 12 months. Patients will be advised to take this medication with food to improve absorption.
  Other Names: Celebrex; Cobix; Celcoxx; Celexib

SUMMARY:
RATIONALE: Celecoxib may stop the growth of thyroid cancer by stopping blood flow to the tumor and by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase II trial to study the effectiveness of celecoxib in treating patients who have progressive metastatic differentiated thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of celecoxib, in terms of progression-free survival, in patients with progressive metastatic differentiated thyroid carcinoma.
* Correlate cyclooxygenase (COX)-2 protein expression in tumor biopsies by immunohistochemistry with clinical response in patients treated with this drug.

OUTLINE: Patients receive oral celecoxib twice daily beginning on day 1. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 3 additional months of therapy beyond documentation of CR.

Patients are followed at 4-8 weeks.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study within approximately 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed thyroid carcinoma, including 1 of the following subtypes:

  * Papillary
  * Follicular
  * Hurthle cell
  * Insular
* Assessable disease, defined by at least 1 of the following:

  * Metastatic (including neck lymph nodes) measurable disease

    * At least 20 mm by conventional techniques or at least 10 mm by spiral CT scan
    * The following are not considered measurable disease:

      * Leptomeningeal disease
      * Ascites
      * Pleural/pericardial effusion
      * Lymphangitis cutis/pulmonis
      * Abdominal masses that are not confirmed and followed by imaging techniques
      * Cystic lesions
      * Tumor lesions within a previously irradiated area
  * Elevated serum thyroglobulin levels indicating the presence of metastatic disease

    * Must have negative thyroglobulin antibodies
* Must have progressive disease within the past year, defined by at least 1 of the following:

  * At least 20% increase in serum thyroglobulin levels
  * At least 20% increase in the sum of the longest diameter of measurable lesions
  * Appearance of at least 1 new lesion
* Failed or ineligible for standard therapy with iodine I 131 and/or surgery

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 1 year

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* AST/ALT no greater than 2 times upper limit of normal

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled cardiac arrhythmia

Gastrointestinal

* No prior symptomatic or complicated peptic ulcer disease by endoscopy within the past 6 months, defined by any of the following conditions:

  * Active gastric or duodenal ulcer
  * Gastric or duodenal perforation
  * Upper gastrointestinal bleeding

Other

* Not pregnant or nursing
* Negative pregnancy test
* No prior allergic reaction to celecoxib or sulfonamides
* No prior urticaria, asthma, or allergic reaction to aspirin or other nonsteroidal anti-inflammatory agents
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled concurrent illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 1 month since prior systemic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 3 months since prior external beam radiotherapy (unless an indicator lesion is outside the radiation field)
* More than 6 months since prior iodine I 131 therapy

Surgery

* See Disease Characteristics
* More than 1 month since prior surgery

Other

* More than 2 weeks since prior conventional doses of celecoxib or rofecoxib for osteoarthritis, rheumatoid arthritis, or dysmenorrhea
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent chronic (more than 1 week of therapy) fluconazole therapy
* Concurrent oral or IV bisphosphonates for bony metastases are allowed
* Concurrent low-dose aspirin (no greater than 325 mg/day) for cardiovascular disease is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Examine efficacy of celecoxib in patients with progressive metastatic differentiated thyroid carcinoma by assessing progression free survival. | up to 12 months following treatment

SECONDARY OUTCOMES:
Quantifying gene expression and protein levels of angiogenic markers[vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), and tumor necrosis factor (TNF)-α] in peripheral blood mononuclear cells (PBMCs) from pre-,during- | pre-study, every eight weeks and off study
Quantifying gene expression and protein levels of cytokines [interleukin (IL)-10, IL-12, IL-6 and interferon (IFN)-γ] in peripheral blood mononuclear cells from pre-,during-, and post-treatment blood samples.
Evaluate cyclooxygenase (COX)-2 protein expression by immunohistochemistry in tumor biopsies to correlate with clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha H. Shah, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comrehensive Cancer Center, Columbus, Ohio
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Mrozek E, Kloos RT, Ringel MD, Kresty L, Snider P, Arbogast D, Kies M, Munden R, Busaidy N, Klein MJ, Sherman SI, Shah MH. Phase II study of celecoxib in metastatic differentiated thyroid carcinoma. J Clin Endocrinol Metab. 2006 Jun;91(6):2201-4. doi: 10.1210/jc.2005-2498. Epub 2006 Mar 7. PMID 16522694
- See also: Jamesline — http://cancer.osu.edu